CLINICAL TRIAL: NCT06329609
Title: Validating the Accuracy of the Airvo 3 Device for Continuous Respiratory Rate Monitoring in Healthy Adults and Chronic Obstructive Pulmonary Disease (COPD) Patients: Comparison With a Reference Benchmark
Brief Title: Airvo 3 Respiratory Rate Validation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ClA-333
Record Dates: First submitted 2024-03-14; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: COPD; Healthy Volunteers
Keywords: High flow therapy; Respiratory rate monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): This arm will receive the study intervention
  Interventions: Device: Airvo 3 with respiratory rate algorithm

INTERVENTIONS:
Device: Airvo 3 with respiratory rate algorithm — Airvo 3 with respiratory rate algorithm is an active humidification system used to deliver high flow respiratory gases (air and/or oxygen) and monitor respiratory rate

SUMMARY:
This is a clinical performance testing to validate the accuracy of the Airvo 3 device with respiratory rate algorithm manufactured by Fisher & Paykel Healthcare for continuous respiratory rate monitoring.

DETAILED DESCRIPTION:
The Airvo 3 device is intended to provide high flow warmed and humidified respiratory gases for administration to spontaneously breathing patients in hospitals and sub-acute facilities. The device has recently been updated with a new feature which allows continuous monitoring of patient's respiratory rate during nasal high flow therapy. This study, therefore, aims to validate the accuracy of the respiratory rate output of the Airvo 3 device. The respiratory rate output of the Airvo 3 device will be compared to the respiratory rate output of a gold standard reference device (capnography) in healthy volunteers and COPD patients to determine the level of agreement between the respiratory rate outputs of the two devices. In addition, the respiratory rate output of the Airvo 3 device will be compared to the respiratory rate output of a United States Food and Drug Administration (U.S. FDA) cleared pulse oximeter in healthy volunteers and COPD patients to determine the level of agreement between the respiratory rate outputs of the two devices.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Healthy adults with no known history of respiratory disease
* Ability to provide written informed consent
* Ability to comply with study procedures and duration

Group B

* Out-patient adults with stable COPD: Global Initiative for Chronic Obstructive Lung Disease (GOLD) stages 2 - 4
* Ability to provide written informed consent
* Ability to comply with study procedures and duration

Exclusion Criteria:

* Pregnancy or lactation
* Inability to tolerate nasal prongs
* History of severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, electrocardiogram (ECG) electrodes, or other medical sensors
* Inability to provide consent
* Participants considered to be medically unsuitable to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | Through study completion, an average of 6 months
  Respiratory rate outputs of investigational device and a gold standard reference device (capnography)

SECONDARY OUTCOMES:
Respiratory rate | Through study completion, an average of 6 months
  Respiratory rate outputs of investigational device and a U.S. FDA cleared pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, MSc, BSN, Principal Investigator — Element Boulder
Locations (1):
- Element Boulder, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No